CLINICAL TRIAL: NCT04181372
Title: A Phase II Study of Neoadjuvant Double-drug Chemotherapy With Platinum Plus Anlotinib Hydrochloride in Stage III(N2) Non-small-cell Lung Cancer
Brief Title: A Study of Neoadjuvant Chemotherapy Plus Anlotinib in Stage III(N2) Non-small-cell Lung Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The First Affiliated Hospital of Guangzhou Medical University (Other)
Responsible Party: Principal Investigator, Jiexia Zhang, Clinical Professor, The First Affiliated Hospital of Guangzhou Medical University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NSCLC 001
Record Dates: First submitted 2019-04-17; First posted 2019-11-29 (Actual); Last update posted 2019-11-29 (Actual); Status verified 2019-11

CONDITIONS: Stage III Non-small-cell Lung Cancer
Keywords: Stage III Non-small-cell Lung Cancer; Anlotinib Hydrochloride; Neoadjuvant
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — anlotinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Anlotinib plus Platinum-based chemotherapy (Experimental): 1. Take anlotinib hydrochloride 12mg once daily for two weeks, stop for one week, the program repeats every 21 days for 2 cycles.
  2. Platinum-based chemotherapy regimens for neoadjuvant:(1)Carboplatin was given dosed to an area under the serum concentration-time curve (AUC) of 6 i.v. injection on day 1, paclitaxel was given 150 mg/m^2 i.v. on day 1, every 21 days for 2 cycles.Or(2) Carboplatin was given dosed to an AUC 5 or Cisplatin was given 75 mg/m^2 ,i.v. on day 1, pemetrexed was given 500 mg/m^2 i.v. on day 1 for nonsquamous, every 21 days for 2 cycles.Or(3) Cisplatin was given 75 mg/m^2 i.v. on day 1; docetaxel was given 75 mg/m^2 i.v. on day 1 ,each 21-day cycle for 2 cycles.
  Interventions: Drug: Anlotinib hydrochloride
- platinum-based chemotherapy (Active Comparator): Platinum-based chemotherapy regimens for neoadjuvant:(1)Carboplatin was given dosed to an AUC of 6 i.v. injection on day 1, paclitaxel was given 150 mg/m^2 i.v. on day 1, every 21 days for 2 cycles.Or(2) Carboplatin was given dosed to an AUC 5 or Cisplatin was given 75 mg/m^2 ,i.v. on day 1, pemetrexed was given 500 mg/m^2 i.v. on day 1 for nonsquamous, every 21 days for 2 cycles.Or(3) Cisplatin was given 75 mg/m^2 i.v. on day 1; docetaxel was given 75 mg/m^2 i.v. on day 1 ,each 21-day cycle for 2 cycles.
  Interventions: Drug: platinum-based chemotherapy medicine

INTERVENTIONS:
Drug: Anlotinib hydrochloride — Anlotinib hydrochloride was given 12mg once daily for two weeks, stop for one week, each 3-week cycle for 2 cycles.
  Other Names: AL3818
  Arms: Anlotinib plus Platinum-based chemotherapy
Drug: platinum-based chemotherapy medicine — (1)Carboplatin was given dosed to an AUC of 6 i.v. injection on day 1, paclitaxel was given 150 mg/m^2 i.v. on day 1, every 21 days for 2 cycles.Or(2) Carboplatin was given dosed to an AUC 5 or Cisplatin was given 75 mg/m^2 ,i.v. on day 1, pemetrexed was given 500 mg/m^2 i.v. on day 1 for nonsquamous, every 21 days for 2 cycles.Or(3) Cisplatin was given 75 mg/m^2 i.v. on day 1; docetaxel was given 75 mg/m^2 i.v. on day 1 ,each 21-day cycle for 2 cycles.
  Arms: platinum-based chemotherapy

SUMMARY:
Stage III non-small-cell lung cancer (NSCLC) is seen in a relatively heterogeneous group of patients with ipsilateral mediastinal (N2) lymph node involvement. The relative roles of different treatment modalities are not clear. The purpose of this study is to evaluate the efficacy and safety of neoadjuvant double-drug chemotherapy containing platinum plus anlotinib hydrochloride in patients with stage III(N2) non-small-cell lung cancer.

DETAILED DESCRIPTION:
This is a prospective, open-label, multi-institutional, positive medicine control of equal rank comparative study of neoadjuvant double-drug chemotherapy with platinum plus anlotinib hydrochloride in stage III(N2) non-small-cell lung cancer.The main purpose of this study was to compare the difference in N2 downgrade rate of lymph node and resectability rate between the experimental and control groups, to evaluate the efficacy of anlotinib hydrochloride, and to observe and evaluate its objective response rate(ORR)，Disease-free Survival (DFS)and overall survival(OS).

ELIGIBILITY:
Inclusion Criteria:

1. Age :18 Years to 75 Years (Adult, Older Adult)
2. Pathological diagnosis with Stage III-N2 NSCLC which is clinically resectable and the N2 is diagnosed by either mediastinoscopy,EBUS,PET/CT;
3. EGFR、ALK、ROS1 mutation-negative；Patients with squamous cell carcinoma may not have genetic testing;PD-L1<5%;
4. According to the RECIST 1.1 standard, there is at least one measurable target lesion;
5. ECOG physical score 0-1 points; expected survival time ≥ 3 months;
6. The main organ function meets the following criteria:1)blood routine: absolute value of neutrophils ≥ 1.5 × 109 / L, platelets ≥ 75 × 109 / L, hemoglobin ≥ 80 g / L;2)Blood biochemistry: total bilirubin ≤ 1.5 times the upper limit of normal value, aspartate aminotransferase and alanine aminotransferase ≤ 2.5 times the upper limit of normal value (if liver metastasis, ≤ upper limit of normal value 5 times), serum creatinine ≤ 1.5 times the upper limit of normal;
7. Subjects voluntarily joined the study and signed informed consent, with good adherence and follow-up.

Exclusion Criteria:

1. Stage I, II , IV orNSCLC;
2. Small cell lung cancer (including lung cancer mixed with small cell lung cancer and non-small cell lung cancer);central lung squamous carcinoma along with cavum;
3. Patients with contraindication of chemotherapy
4. Subjects who have previously used Anlotinib;
5. Systematic anti-tumor treatments have been performed for the past 2 weeks, including chemotherapy, radiotherapy (except for metastatic lesions other than thoracic radiation), targeted therapy, immunotherapy, and biotherapy;
6. Imaging (CT or MRI) shows that the distance between tumor lesion and the large blood vessel is ≤ 5 mm, or there is a central tumor that invades the local large blood vessel; or there is a significant pulmonary cavity or necrotizing tumor;
7. A history of active bleeding within the first 6 months of screening, or receiving thrombolysis or anticoagulant therapy, or the investigator believes that there is a clear tendency to gastrointestinal bleeding (such as esophageal varices with bleeding risk, local activity) Ulcer lesions, etc.) or active hemoptysis;
8. A thrombotic event occurs within 6 months (including arteriovenous thrombosis, pulmonary embolism, cerebrovascular accident, including transient ischemic attack, etc.);
9. Cardiac diseases with obvious clinical symptoms, such as: congestive heart failure, coronary heart disease with obvious symptoms, arrhythmia with difficult drug control (including clinically significant QTc interval prolongation history, or screening period QTc interval women >470ms, Male > 450ms), had myocardial infarction within 6 months, or cardiac insufficiency;
10. Hypertension, which is uncontrolled by the drug, is defined as: systolic blood pressure ≥ 160 mmHg, or diastolic blood pressure ≥ 100 mmHg;
11. Clinically obvious gastrointestinal abnormalities, which may affect the intake, transport or absorption of drugs (such as inability to swallow, chronic diarrhea, intestinal obstruction, etc.), or patients with total gastrectomy;
12. Surgery (<28 days) before the study was selected or the surgical incision did not completely heal, or there were other unhealed wounds;
13. Active or uncontrolled serious infections;
14. Pregnant or lactating women; those who have fertility are unwilling or unable to take effective contraceptive measures;
15. Increasing the risk associated with participating in a study or study drug, and at the discretion of the investigator, may lead to other conditions in which the patient is not eligible for inclusion in the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2019-12 (Estimated); Primary Completion 2021-08-01 (Estimated); Study Completion 2022-08-01 (Estimated)

PRIMARY OUTCOMES:
Lymph node(N2)downstage rate | 3 months
  Lymph node downstage rate is depended on the image or pathology dignosis after surgery,staging from N2 to N1 / N0.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | 3 months
  ORR is the number of participants with a Complete Response (CR) and Partial Response (PR) divided by the total number of randomized participants per arm, then multiplied by 100. Response is based on the Response Evaluation Criteria In Solid Tumors (RECIST 1.1) criteria. Complete Response (CR) was defined as the disappearance of all target lesions. Partial Response (PR) was defined as at least a 30% decrease in sum of longest diameter of target lesions compared to baseline or the complete disappearance of target lesions, with persistence of 1 or more nontarget lesion(s) and no new lesions.
Resectability rate | Lymph node downstage rate is depended on the pathology dignosis after surgery, an expected average of 8 weeks from randomization.
  Resectability rate was defined as the percentage of patients who were able to undergo surgery after neoadjuvant therapy.
Pathological complete response (pCR) rate | 3 months
  Pathologic Complete Response Rate is defined as lack of evidence of viable cancer in the surgical specimen at the time of surgery.
Disease-free Survival （DFS） | Every 3 months.
  The period after curative treatment [disease eliminated] when no disease can be detected.From date of randomization until the date of first documented progression, whichever came first, assessed up to 40 months.
Overall Survival (OS) | 3 years
  OS was assessed from randomization to death as a result of any cause.
adverse events(AEs) | 3 months
  Number of participants with perioperative complications.

CONTACTS AND LOCATIONS:
Overall Officials: Jiexia Zhang, prof., Study Chair — The First Affiliated Hospital of Guangzhou Medical University
Locations (1):
- The First Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong, China